CLINICAL TRIAL: NCT06085638
Title: Phase I/II Study of SY-1425 (Tamibarotene) in Combination With Azacitidine and Venetoclax for Patients With Chronic Myelomonocytic Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Zero participants accrued
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Syros Pharmaceuticals Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0110; NCI-2023-08582 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine; tamibarotene; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm1: Cohort 1: Azacitidine + Tamibarotene (Experimental): Participants will receive azacitidine on Days 1-7 of each cycle and tamibarotene 2 times a day every day. Up to 20 participants will be enrolled in Cohort 1.
  Interventions: Drug: Azacitidine; Drug: Tamibarotene
- Arm2: Cohort 2,3: Azacitidine + Tamibarotene + Venetoclax (Experimental): Participants will receive azacitidine on Days 1-7 of each cycle, tamibarotene 2 times a day every day, and venetoclax on either Days 1-7 or Days 1-14 of each cycle, depending on the dose level you are assigned at enrollment. Up to 12 participants will be enrolled in Cohort 2.
  Once Cohort 2 is complete, Cohort 3 will begin. Participants in Cohort 3 will receive the recommended dosing schedule found in Cohort 2 (azacitidine on Days 1-7, tamibarotene 2 times a day every day, and venetoclax on either Days 1-7 or Days 1-14
  Interventions: Drug: Azacitidine; Drug: Tamibarotene; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given by SC (under the skin) or IV (vein)
  Other Names: 5-azacytidine; 5-aza; Vidaza™; 5-AZC; AZA-CR; Ladakamycin; NSC-10281
Drug: Tamibarotene — Given by PO
Drug: Venetoclax — Given by PO
  TAMIBAROTENE Azacitidine Azacitidine, 5-azacytidine, 5-aza, Vidaza™, 5-AZC, AZA-CR, Ladakamycin, NSC-102816, Azacytidine Venetoclax ABT-199, GDC-0199, Venetoclax
  Other Names: ABT-199; GDC-0199
  Arms: Arm2: Cohort 2,3: Azacitidine + Tamibarotene + Venetoclax

SUMMARY:
To learn if adding venetoclax to the chemotherapy combination of tamibarotene and azacitidine is more effective than tamibarotene and azacitidine alone in treating higher-risk CMM

DETAILED DESCRIPTION:
Primary Objectives:

* Cohort 1: Characterize the safety and toleratbility of the combination of azacitidine and tamibarotene in newly diagnosed CMML.
* Cohort 2 and 3: Characterize the safety and tolerability of tamibarotene in combination with azacitidine and venetoclax in relapsed higher risk CMML.

Secondary Objectives:

* Cohort 1: Characterize the preliminary clinical activity of tamibarotene in combination with azacitidine defined by complete response (CR) rate, following MDS/MPN IWG response criteria (Appendix 1),
* Cohort 2: Characterize the safety and tolerability of tamibarotene in combination with azacitidine and venetoclax in relapsed higher risk CMML.
* Cohort 3: Characterize the clinical activity of tamibarotene in combination with azacitidine and venetoclax by overall response rate (ORR) in relapsed higher risk CMML.
* To characterize additional clinical activity outcomes such as duration of response, leukemia-free survival (LFS), event-free survival (EFS) and overall survival (OS).
* To evaluate differences in response and efficacy outcomes by MDS/MPN IWG response criteria based on RARA expression levels and positivity.
* To correlate response with disease subtype and genomic profile
* To evaluate changes in clonal composition and VAF of identified mutations with therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years old
2. CMML according to WHO and:

   Cohort 1: HMA-naïve CMML-2 or HMA-naïve CMML-1, with Int-1, Int-2 or high risk by the Molecular CMML-Specific Prognostic Scoring system (CPSS-Mol) in whom HMA therapy is indicated.

   Cohorts 2 and 3: CMML-1 or CMML-2 and failure to HMA defined as no response after 4 cycles of azacitidine, decitabine, guadecitabine, oral decitabine/cedazuridine, ASTX030, or relapse or progression after any number cycles.
3. ECOG Performance Status of ≤2.
4. Patients must have the following laboratory values:

   total bilirubin ≤1.5 × the ULN (Patients with Gilbert's syndrome can be included with total bilirubin >1.5 x ULN as long as direct bilirubin is < 35% of total bilirubin and ≤ 1.5 x ULN) ALT and AST ≤2.5 × ULN, and creatinine clearance ≥60 mL/min based on the Cockcroft-Gault Glomerular Filtration Rate estimation.
5. Patients must have a serum or high-sensitivity urine pregnancy test (for females of childbearing potential) that is negative at the Screening Visit and within 72 hrs prior to initiation of treatment (first dose of study drug).
6. Patients must be willing and able to comply with the scheduled study visits, treatment plans, laboratory tests, use of 2 methods of birth control (including a barrier method) for patients who are women of childbearing potential (WOCBP) and for male patients
7. White blood cell (WBC) count <50,000/L (<10,000/L prior to starting Cycle 1 Day 1 with venetoclax on Cohorts 2 and 3). Hydroxyurea may be used to control leukocytosis prior to and for the first 28 days of study treatment (i.e cycle 1). Use of hydroxyurea beyond this point may be permitted as clinically indicated, on a case-by-case basis and after discussion with the PI.

Exclusion Criteria:

1. Patients who are currently receiving treatment for a malignancy (not including basal cell carcinoma, non melanoma skin cancer, cervical carcinoma in situ, or localized prostate cancer treated with hormone therapy). Patients with history of other cancers should be free of disease for at least 2 years prior to the Screening Visit.
2. Patients who have an active, life-threatening, or clinically-significant uncontrolled systemic infection requiring hospitalization.
3. Patients who have a known malabsorption syndrome or other condition that may impair absorption of study medication (e.g., gastrectomy).
4. Immunocompromised patients with increased risk of opportunistic infections, including known HIV-positive patients with CD4 counts ≤350 cells/mm3 or history of opportunistic infection in the last 12 months. Note: To ensure that effective ART, when used in eligible HIV-positive patients, is tolerated and that toxicities are not confused with investigational drug toxicities, patients should be on an established ART for at least 4 weeks and have an HIV viral load less than 400 copies/mL prior to the Screening Visit.
5. Patients with a known active or chronic hepatitis B or active HCV infection. Patients with a history of HCV infection who have completed curative therapy for HCV at least 12 weeks before the Screening Visit and have a documented undetectable viral load at the Screening Visit are eligible for enrollment.
6. Patients who have other severe acute or chronic medical conditions (and/or psychiatric conditions or laboratory abnormalities) that may increase the expected risk to the patient (i.e., the risk associated with the study participation or study drug administration) or that may interfere with the interpretation of study results or, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
7. Patients who have not adequately recovered from a major surgery within 4 weeks prior to starting study drug administration.
8. Patients with a diagnosis of hypervitaminosis A or patients taking vitamin A supplements >10,000 IU/day, unless treatment is discontinued at least 7 days prior to the first dose of the study drug.
9. Patients received strong inducers of CYP3A4 (see Appendix 4) within 2 weeks prior to the first tamibarotene administration.
10. Patients who received any other investigational agents within 4 weeks prior to the Screening Visit or <5 half-lives since completion of previous investigational therapy have elapsed, whichever is shorter.
11. Patients require concurrent treatment with any investigational or approved oncology agent.
12. Patients with Grade ≥2 hypertriglyceridemia, defined as >300 mg/dL (CTCAE, version 5).
13. Patients with QTc interval >480 msec based on average of triplicate ECG readings at the Screening Visit using the Fridericia formula (QTcF), with the exception of patients with right bundle branch block or left bundle branch block.
14. Pregnant females, breastfeeding females, and males or females of childbearing potential not willing to comply with contraceptive requirements (as described in Appendix 2)
15. Patients who have a hypersensitivity to tamibarotene, azacitidine or venetoclax, or to any of their excipients, including sodium hydrosulfite.
16. Patients for whom treatment with tamibarotene is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Montalban Bravo, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org